CLINICAL TRIAL: NCT00966732
Title: Yoga of Awareness Program for Fibromyalgia: A Randomized Clinical Trial
Brief Title: Yoga for Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, James W Carson, PhD, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Yoga for Fibromyalgia
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- yoga condition (Experimental): assigned to start the yoga program right away
  Interventions: Behavioral: Yoga of Awareness Program
- wait-list control condition (No Intervention): This condition will control for any effects of symptom measurement reactivity in patients receiving routine fibromyalgia medical care. After the 3-month assessment, the yoga intervention program will be provided to these patients.

INTERVENTIONS:
Behavioral: Yoga of Awareness Program — The 8 week yoga program will meet in groups of about 8-10 persons. Each 2-hour session will include gentle stretching, strengthening, and balance poses; meditation exercises; breathing techniques; study of pertinent topics (eg, mind/body stress reactivity), and group discussions (eg, experiences while practicing yoga). Participants will be asked to practice yoga methods at home, guided by a DVD (or audio recordings). The program will be taught by a certified yoga teacher (RYT) who has extensive experience in teaching yoga to medical patients.
  Arms: yoga condition

SUMMARY:
Fibromyalgia is a common, costly and debilitating illness which affects mostly women. Fibromyalgia patients report widespread musculoskeletal pain, fatigue, stiffness, and distress. Several consensus statements indicate that optimal care combines medication, exercise, and psychology. Yoga is a popular mind/body discipline which holds promise for reducing fibromyalgia symptoms. The aim of this pilot study is to evaluate the effects of an innovative program, Yoga of Awareness, in which yoga poses are complemented by meditation and breathing exercises, presentations on healthy coping, and group discussions. Fifty-six women with fibromyalgia will be recruited and randomly divided into two groups. One group will receive the yoga program right away, and the other group will wait 3 months before receiving the program. Information about fibromyalgia symptoms and functioning will be collected from both groups before and immediately after the first group receives the yoga program. When results from the 2 groups are compared, the investigators expect patients who received the yoga program will have greater gains in fibromyalgia symptoms, physical function and pain coping capacities then those waiting to receive the program. If this study shows the yoga program is effective, the investigators will use this data in 2010 to apply to the National Institutes of Health for a more complete study of its benefits.

ELIGIBILITY:
Inclusion Criteria:

* women ≥21 years of age
* diagnosed with fibromyalgia by ACR criteria for at least 1 year
* on a stable regimen of pharmacologic and/or non-pharmacologic treatment for FM ≥3 months

Exclusion Criteria:

* reside >70 miles from the research site
* unavailable to attend the intervention at one of the scheduled times
* currently engaged in intensive yoga practice (practice >3 days/wk)
* score >29 on the Beck depression scale modified for fibromyalgia
* currently undergoing disability application or involved in litigation
* elective surgery scheduled during the study period
* physically disabled in a manner that precludes meaningful participation in the intervention (eg, quadriplegic paralysis)
* do not speak English

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2009-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire Revised (FIQR) | baseline, 3 months, 6 months

SECONDARY OUTCOMES:
Vanderbilt Multidimensional Pain Coping Inventory (VMPCI) | baseline, 3 months, 6 months
Chronic Pain Acceptance Questionnaire (CPAQ) | baseline, 3 months, 6 months
Coping Strategies Questionnaire Catastrophizing Subscale (CSQCAT) | baseline, 3 months, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: James W Carson, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States